CLINICAL TRIAL: NCT04346901
Title: Comparative Study of mMASI Before and After Hyperthyroid Therapy in Hyperthyroid Subjects With Melasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Irma Bernadette S. Sitohang, MD, PhD - Head of Division of Cosmetic Dermatology, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TesBN
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Melasma; Hyperthyroidism
Keywords: Melasma; modified melasma area and severity index; Thyroid stimulating hormone; Free thyroxine
MeSH Terms: conditions — Melanosis; Hyperthyroidism | interventions — Methimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Intervention (Other): Before-and-After type of research
  Interventions: Drug: Thiamazol

INTERVENTIONS:
Drug: Thiamazol — All new hyperthyroid with melasma patients were recruited and their mMASI were calculated All subjects were given thiamazole by Internist based on their clinical hyperthyroidism After 3 months of taking hyperthyroid drugs (thiamazole), mMASI were recalculated and compared

SUMMARY:
Study's objectives are to determine proportion of melasma cases in hyperthyroid patients and to compare severity of melasma before and after medications of three months hyperthyroid therapy using modified melasma area and severity index (mMASI) score. A quasi experimental (pre-post intervention) study was conducted in Jakarta in August 2019-February 2020.

DETAILED DESCRIPTION:
Melasma is an acquired and chronic disorder of hyperpigmentation characterized by symmetrical hypermelanoses of the face. The exact pathogenesis of melasma is still unknown. Several hormones are thought to play a role, including thyroid hormone. Although melasma is not life-threatening, it affects greatly on the quality of life of patients. Study's objectives are to determine proportion of melasma cases in hyperthyroid patients and to compare severity of melasma before and after medications of three months hyperthyroid therapy using mMASI score. An experimental (before and after) study was conducted in Jakarta in August 2019-February 2020. Twenty three newly-diagnosed hyperthyroid patients or had taken hyperthyroid medications of maximum 3 months with melasma were recruited. The severity of melasma were scored with mMASI and dermoscopy of the lesions were collected. The same procedures were done after 3 months of hyperthyroid therapy. The data collected was statistically analyzed using Stata version 15.0

ELIGIBILITY:
Inclusion Criteria:

* Female with age range of 18 to 60 years old
* Newly diagnosed with hyperthyroid on a laboratory basis
* Diagnosed with melasma by dermatologist

Exclusion Criteria:

* Pregnant or breastfeeding
* Using hormonal contraception or history of using hormonal contraception within 1 year
* On anti-seizure therapy or hormone replacement therapy
* History of drug use that can affect the thyroid
* History of using topical hydroquinone in the last 3 months and / or using a topical steroid and / or an vitamin A analog and / or received chemical peeling in the last 1 month
* History of laser therapy and / or mechanical abrasion therapy in the past 9 months

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
mMASI (modified melasma area and severity index) | 3 months after taking the hyperthyroid drugs
  mMASI Score (modified melasma area and severity index); value 0-24; smaller score means better outcome

OTHER OUTCOMES:
Proportion of melasma in hyperthyroid patients | 3 months
  Melasma proportion in hyperthyroid patients who visited the policlinics

CONTACTS AND LOCATIONS:
Overall Officials: Irma B Sitohang, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- dr. Cipto Mangunkusumo Hospital, Jakarta, Jakarta Pusat, Indonesia